CLINICAL TRIAL: NCT07315542
Title: Finding New Diagnostic and Therapeutic Targets in Cartilaginous Tumours
Brief Title: Diagnostic and Therapeutic Targets in Cartilaginous Tumours
Status: Recruiting | Type: Observational
Sponsor: St. Anne's University Hospital Brno, Czech Republic (Other)
Collaborators: Masaryk University (Other)
Responsible Party: Sponsor
Other Study IDs: NW25-10-00260; NW25-10-00260 (Other Grant/Funding Number: Ministry of Health Research Programme 2024 - 2030)
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Chondrosarcomas; Cartilage Tumours
Keywords: Chondrosarcoma; Liquid biopsy; Targeted therapy; Prognostic markers; Molecular biomarkers; MicroRNA (miRNA); Cartilaginous tumours; IDH1 mutation; IDH2 mutation
MeSH Terms: conditions — Chondrosarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — tumor samples blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with cartilaginous bone tumours: The study cohort consists of patients with cartilaginous bone tumours treated at a tertiary orthopaedic oncology centre. This includes individuals with benign, borderline, and malignant chondroid lesions across the full biological spectrum, namely enchondromas, atypical cartilaginous tumours (ACT/G1), conventional chondrosarcomas (grades G1-G3), dedifferentiated chondrosarcomas, and selected rare variants. Interventions of interest in this study are primarily diagnostic and molecular, rather than therapeutic in the interventional trial sense.
  Molecular analysis of tumour tissue using next-generation sequencing (NGS) to assess global microRNA expression profiles and IDH1/2 mutation status.
  Validation of selected molecular markers using RT-qPCR and targeted mutation detection assays. Analysis of circulating and exosomal microRNAs from blood as a form of liquid biopsy. Experimental miRNA modulation to investigate biological relevance in relation to IDH1/2 mutation status.
  Interventions: Diagnostic Test: Tumour tissue analysis; Diagnostic Test: Molecular validation; Diagnostic Test: Liquid biopsy analysis

INTERVENTIONS:
Diagnostic Test: Tumour tissue analysis — Next-generation sequencing (NGS) to determine IDH1/2 mutation status
  Global microRNA (miRNA) expression profiling using NGS
Diagnostic Test: Molecular validation — Quantitative reverse transcription PCR (RT-qPCR) to validate selected miRNAs
  Targeted molecular assays for confirmation of IDH1/2 mutations
Diagnostic Test: Liquid biopsy analysis — Assessment of circulating and exosomal miRNAs from patient body fluids as non-invasive biomarkers

SUMMARY:
This study, "Finding new diagnostic and therapeutic targets in cartilaginous tumours," focuses on improving the diagnosis, prognostic stratification, and treatment options for chondroid tumours, particularly chondrosarcoma. Chondrosarcoma is the most common primary malignant bone tumour in adults and is characterized by resistance to chemotherapy and radiotherapy, making accurate diagnosis and optimal surgical management critical. Distinguishing benign cartilage tumours (enchondromas, atypical cartilaginous tumours) from low-grade chondrosarcoma, and differentiating chondrosarcoma from chondroblastic osteosarcoma, remain major diagnostic challenges.

The project investigates two key molecular markers: mutations in IDH1/2 genes and non-coding microRNAs (miRNAs). IDH1/2 mutations are frequent in central chondrosarcomas and rare in other mesenchymal tumours, making them promising diagnostic markers. Their presence may also have prognostic significance and therapeutic relevance, as IDH inhibitors are already available for other malignancies. In parallel, deregulated miRNA expression has been implicated in chondrosarcoma biology, influencing tumour growth, invasion, angiogenesis, metastasis, and chemosensitivity. Preliminary data identified distinct miRNA signatures in chondrosarcoma compared with healthy cartilage, including previously unreported miRNAs.

The study is structured into exploratory and validation phases. Global miRNA expression profiling and IDH1/2 mutation analysis will be performed using next-generation sequencing (NGS) on prospectively collected fresh-frozen tumour samples. Selected miRNAs and IDH1/2 mutation status will then be validated by RT-qPCR and targeted mutation assays in a large retrospective cohort of FFPE samples. Molecular data will be integrated with clinicopathological parameters to develop diagnostic panels capable of accurately classifying chondroid tumours, as well as prognostic miRNA panels associated with patient survival.

Additionally, the project evaluates circulating and exosomal miRNAs in liquid biopsies, aiming to establish non-invasive diagnostic and prognostic tools. Functional relevance will be explored using chondrosarcoma cell lines with simulated miRNA upregulation, coupled with transcriptomic analysis.

Overall, the study seeks to refine diagnostic accuracy, improve prognostic assessment, and identify novel molecular targets for personalized and targeted therapy in patients with inoperable or metastatic chondrosarcoma, addressing a major unmet clinical need.

DETAILED DESCRIPTION:
The study entitled "Finding new diagnostic and therapeutic targets in cartilaginous tumours" addresses major unresolved problems in the diagnosis, prognostic assessment, and treatment of chondroid tumours, with a particular focus on chondrosarcoma. Chondrosarcoma represents approximately 30% of all primary malignant bone tumours and is the most common malignant bone sarcoma in adults. Despite its clinical relevance, the management of chondrosarcoma remains challenging due to its biological heterogeneity, resistance to chemotherapy and radiotherapy, and frequent diagnostic uncertainty, especially in low-grade lesions.

A central clinical problem lies in the differentiation between benign cartilage tumours (enchondromas and atypical cartilaginous tumours), low-grade chondrosarcoma, higher-grade chondrosarcoma, and other malignant entities such as chondroblastic osteosarcoma. Histological assessment alone is often insufficient, particularly in small biopsy specimens, and diagnostic decisions frequently rely on a subjective combination of clinical, radiological, and pathological criteria. Incorrect classification may lead either to undertreatment with insufficient local control or overtreatment with unnecessarily radical surgery. Furthermore, advanced, inoperable, or metastatic chondrosarcoma has a very poor prognosis, and effective systemic therapies are currently lacking.

This project focuses on the identification and validation of molecular biomarkers that could significantly improve diagnostic precision, prognostic stratification, and therapeutic targeting. Two main molecular areas are investigated: IDH1/2 gene mutations and non-coding microRNAs (miRNAs).

Mutations in IDH1 and IDH2 genes have been identified as characteristic molecular events in cartilaginous tumours. These mutations occur at specific amino acid residues and lead to neomorphic enzymatic activity, resulting in the production of the oncometabolite 2-hydroxyglutarate. IDH1/2 mutations are common in central chondrosarcomas and related benign precursors but are rare or absent in peripheral chondrosarcomas and other mesenchymal tumours, including osteosarcoma. As such, IDH1/2 mutation status represents a highly valuable diagnostic marker, particularly for distinguishing chondrosarcoma from chondroblastic osteosarcoma, a distinction with major therapeutic implications. The study also hypothesizes that IDH1/2 mutations may be associated with tumour aggressiveness and poorer prognosis, making them potential prognostic markers and therapeutic targets. Importantly, IDH inhibitors already used in other malignancies may represent a future treatment option for selected chondrosarcoma patients.

The second major focus of the project is the role of microRNAs, short non-coding RNAs that regulate gene expression at the post-transcriptional level. Numerous studies have shown that miRNA dysregulation contributes to tumour initiation, progression, angiogenesis, invasion, and metastasis. In chondrosarcoma, specific miRNAs have been implicated in the regulation of key oncogenic pathways, including SRC, mTOR, Wnt/β-catenin signalling, VEGF-mediated angiogenesis, and matrix remodelling. Preliminary next-generation sequencing data generated by the research team identified distinct miRNA expression profiles in chondrosarcoma compared with healthy cartilage, including several miRNAs not previously reported in the literature. These findings support the existence of tumour-specific miRNA signatures with diagnostic and prognostic potential.

The study is designed in exploratory and validation phases. In the exploratory phase, prospectively collected fresh-frozen tumour samples will undergo global miRNA expression profiling using next-generation sequencing, alongside NGS-based analysis of IDH1/2 mutation status. This phase aims to identify characteristic molecular patterns across the spectrum of chondroid tumours, including benign lesions, low-grade and high-grade chondrosarcoma, dedifferentiated variants, and chondroblastic osteosarcoma.

In the validation phase, selected deregulated miRNAs and IDH1/2 mutations will be analysed in a large retrospective cohort of FFPE samples using RT-qPCR and targeted mutation detection methods. Molecular results will be integrated with detailed clinicopathological data to develop robust diagnostic miRNA panels capable of accurately classifying chondroid tumours and distinguishing chondrosarcoma from osteosarcoma. In parallel, prognostic miRNA panels will be established and correlated with overall survival using advanced statistical methods, including Kaplan-Meier analysis and Cox proportional hazards modelling.

An innovative component of the project is the evaluation of liquid biopsies, analysing circulating and exosomal miRNAs from patient body fluids. This approach aims to establish non-invasive biomarkers for diagnosis, prognosis, and disease monitoring beyond the time of surgery. Additionally, functional relevance will be explored using chondrosarcoma cell lines, in which selected miRNAs will be experimentally upregulated to assess downstream transcriptomic effects and their relationship to IDH1/2 mutation status.

Overall, this study aims to significantly advance the understanding of chondrosarcoma biology and translate molecular findings into clinically applicable tools. By improving diagnostic accuracy, enabling prognostic stratification, and identifying novel therapeutic targets, the project addresses a critical unmet need in the management of cartilaginous tumours and lays the groundwork for future targeted and personalized treatment strategies.

ELIGIBILITY:
Inclusion Criteria

* Histologically confirmed cartilaginous (chondroid) tumour
* Diagnosis includes one of the following entities (as available and eligible):
* Enchondroma
* Atypical cartilaginous tumour / Grade 1 chondrosarcoma (ACT/G1)
* Conventional chondrosarcoma (Grade 2-3)
* Dedifferentiated chondrosarcoma
* Other rare chondrosarcoma variants (e.g., mesenchymal, clear-cell), if present in the cohort
* Patients treated and/or followed at the First Department of Orthopaedic Surgery, St. Anne's University Hospital Brno

Exclusion Criteria

* Insufficient, degraded, or otherwise unusable tissue samples

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of patients with cartilaginous (chondroid) tumours treated at the First Department of Orthopaedic Surgery, St. Anne's University Hospital Brno, a national referral centre for bone tumours.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of molecular markers | From May 2025 to December 2027
  Ability of IDH1/2 mutation status and tumour tissue miRNA expression profiles to: Distinguish benign cartilaginous tumours (enchondromas, atypical cartilaginous tumours) from malignant tumours (chondrosarcomas). Distinguish chondrosarcoma from chondroblastic osteosarcoma. Outcomes will be quantified using molecular classification performance (e.g. correct stratification against histopathological diagnosis) based on NGS and RT-qPCR analyses.
Identification of prognostic molecular signatures | From May 2025 to December 2027
  Association between IDH1/2 mutation status and overall survival of patients with malignant cartilaginous tumours.
  Identification of prognostic miRNA panels whose expression profiles stratify patients into different survival risk groups.

SECONDARY OUTCOMES:
Validation of candidate biomarkers | From May 2025 to December 2027
  Technical and biological validation of selected deregulated miRNAs and IDH1/2 mutations in an independent retrospective FFPE cohort using RT-qPCR and targeted mutation assays.
  Reproducibility and stability of miRNA panels across different sample types (fresh-frozen vs FFPE tissue).
Liquid biopsy feasibility | From May 2025 to December 2027
  Detection and quantification of circulating and exosomal miRNAs in prospectively collected body fluids.
  Concordance between miRNA profiles in liquid biopsies and matched tumour tissue samples.

CONTACTS AND LOCATIONS:
Overall Officials: Tomáš Tomáš, Assoc.Prof., M.D., Ph.D., Principal Investigator — Faculty of Medicine, Masaryk University, Brno, 60200, Czechia; Michal Mahdal, M.D., Ph.D., Principal Investigator — First Department of Orthopaedic Surgery, St. Anne's University Hospital, Brno, 60200, Czechia
Locations (1):
- First Department of Orthopaedic Surgery, St. Anne's University Hospital and Faculty of Medicine, Masaryk University, Brno, Czechia, Brno, South Moravian, Czechia

IPD SHARING:
Plan to Share IPD: No